CLINICAL TRIAL: NCT00964964
Title: A Trial Assessing the Number of Hypoglycaemic Episodes and Glycaemic Variability During Two Different Regimens of SIBA 200 U/ml in Subjects With Type 1 Diabetes
Brief Title: A Trial Assessing Changes in Blood Sugar and the Number of Periods Where Supplementation of Carbohydrate is Needed to Treat Low Blood Sugar, During Two Different Treatment Regimens of NN1250 in Type 1 Diabetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1250-3765; 2009-011959-53 (EudraCT Number)
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIBA 3W (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- SIBA OD (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Insulin degludec injected s.c. (under the skin) three times weekly
  Arms: SIBA 3W
Drug: insulin degludec — Insulin degludec injected s.c. (under the skin) once daily for one week
  Arms: SIBA OD
Drug: placebo — Placebo injected s.c. (under the skin) four times weekly
  Arms: SIBA 3W

SUMMARY:
This trial is conducted in Europe. The aim is to compare changes in blood sugar and the number of periods where carbohydrate supplementation is needed to treat low blood sugar, during two different treatments with NN1250 (insulin degludec), a soluble insulin basal analogue (SIBA) in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months
* Glycosylated haemoglobin (HbA1c) between 7.5 and 9% (both inclusive)

Exclusion Criteria:

* Donation or loss of more than 500 ml blood or plasma within three months prior to this trial
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day) or not able or willing to refrain from smoking and the use of nicotine gum or transdermal nicotine patches during the in-house periods
* Prior or current treatment with metformin or thiazolidinediones

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Total number of periods where carbohydrate supplementation is needed during the treatment | Assessed every day of the two in-house stays of nine days

SECONDARY OUTCOMES:
Frequency of adverse events (AEs) | Assessed every day of the two in-house stays of nine days and one follow-up by telephone
Number of periods with low blood sugar during treatment | Assessed every day of the two in-house stays of nine days and one follow-up by telephone

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com